CLINICAL TRIAL: NCT06266468
Title: Nutricity: An mHealth Nutrition Intervention to Improve Diet Quality Among Latino Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00149178
Record Dates: First submitted 2024-01-11; First posted 2024-02-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Diet Quality

STUDY DESIGN:
Intervention Model Description: The intervention study model is a 2-arm randomized control trial with a 1:1 allocation of participants to the treatment group (Nutricity) or the control group (usual care without Nutricity). After 12 weeks in the control group, participants will be introduced to Nutricity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 12 weeks of mobile intervention (website and text messaging)
  Interventions: Behavioral: Nutricity
- Waitlist (Placebo Comparator): No intervention for 12 weeks, or until completion of 2nd study visit
  Interventions: Behavioral: Nutricity

INTERVENTIONS:
Behavioral: Nutricity — Nutricity is a bilingual (English/Spanish) mobile website supplemented by an automated text-messaging system.

SUMMARY:
The overall objective of this application is to pilot test an mHealth nutrition intervention within pediatric clinics serving Latino families and evaluate its potential for implementation. The investigators hypothesize the intervention will improve child diet quality and will be feasible for use within the clinic setting. To test this hypothesis, the investigators will pursue 3 specific aims and 1 exploratory aim:

1. Aim 1: Pilot Nutricity with 40 Latino families (English or Spanish speaking) vs. 40 waitlist control in primary care clinics and estimate differences in child diet quality at 3 month's post Nutricity exposure. Preliminary data will inform power calculations for a future larger Nutricity intervention.
2. Aim 2: Evaluate other individual (dyad) level factors including reach, engagement, and changes in secondary effectiveness outcomes (e.g. nutrition literacy, BMI, skin carotenoid, psychosocial constructs) at 3 months post exposure.
3. Aim 3: Evaluate organizational-level factors (adoption, implementation, and organizational-level maintenance) in Latino-serving pediatric clinics that may support or inhibit future uptake of Nutricity. The investigators will seek to understand the context of interventions and scalability to other clinics using mixed methods.
4. Exploratory Aim 1: Explore the relationship among nutrition literacy, psychosocial constructs and diet quality outcomes; and explore how engagement and satisfaction influence outcomes.

DETAILED DESCRIPTION:
There are three phases of participation in this study:

Phase 1 (Baseline): Participating parent and child dyads will be asked to come to the clinic or research lab 1 time for procedures and assessments that will help the investigator assess nutrition knowledge and eligibility. Assessment collected at this time will include: 1) Height/Weight: Parent and child will have their height and weight measured; 2) Demographics: survey with questions including items such as name, date of birth and race; 3)Two Nutrition Questionnaires: Nutrition Literacy Assessment Instrument (NLit, measures nutrition knowledge of nutrition and health, energy sources in food, household food measurement, food labels/numbers, food groups and consumer skills) and a food intake screening survey; 4)24-hour Recall: Parents will be asked questions about their child's current diet over the last 24 hours. For children who eat meals at school or daycare, researchers may ask parents to provide forms for the child's teacher or daycare provider to record the meals they eat while there. Parents will also be asked to do two additional recall during the study that will be done with researchers over the phone; 5)Resonance Raman Spectroscopy (Veggie Meter): During this assessment, the veggie meter will apply gentle pressure to the pad of the child's fingertip to put it in close contact with light, to detect and measure carotenoid in the blood. Three, 10-45 second measurements are taken and averaged for the recorded score. Phase 2 (Nutricity): During this phase participants will use their smartphone or tablet to access the Nutricity website to potentially increase nutrition literacy and set nutrition goals by text message. Participants will have their own user name and password to access the site. This phase will last approximately 3 months. Phase 3 (End Study): Participant dyads will be asked to come to the research lab 1 time to perform the same procedures and assessments completed in the baseline visit as well as one exit survey.

ELIGIBILITY:
Inclusion Criteria:

* Age (of parent) > 18 years;
* Parent or guardian of a child between 1-5 years old;
* Hispanic/Latino;
* English or Spanish speaking;
* Primary food decision-maker for the home;
* Internet connectivity at home (smart phone is adequate);
* Owns a device for accessing internet at home.

Exclusion Criteria:

* Overt cognitive or psychiatric illness;
* Visual impairments that preclude viewing educational materials and using a tablet/device;
* Child illness requiring a highly restrictive diet, such as type 1 diabetes, renal disease, celiac disease, etc.;
* Another parent/guardian-child dyad in the household is enrolled in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Diet quality (Healthy Eating Index) (child) | Baseline and at 3 months
  Healthy Eating Index (HEI) calculated from nutrient data derived from 2, 24-hour recalls. Healthy Eating Index (HEI) scores range from 0 to 100. A score of 100 means a better outcome, reflecting that foods align with key dietary recommendations and dietary patterns published in the Dietary Guidelines.

SECONDARY OUTCOMES:
Nutrition Literacy (parent) | Baseline and at 3 months
  Measured by the Nutrition Literacy Assessment Instrument (score ranges 0 to 42). Scores are interpreted as: >39 good, 29-38: moderate, ≤ 28: poor.
Body Mass Index (child) | Baseline and at 3 months
  Calculated from measured height and weight. Body Mass Index can range from ≤18.5 to ≥30. A Body Mass Index between 18.5 and 24.9 is within the Healthy Weight range.
Skin Carotenoid | Baseline and at 3 months
  Assesses carotenoid status, a biomarker of fruit and vegetable intake. Scale ranges between 0 and 800. A higher score means a better outcome.
Feeding Behaviors of Parent and Children | Baseline and at 3 months
  Behavioral Pediatrics Feeding Assessment Scale (BPFAS): A 35-item parent report of child mealtime and feeding behaviors- this scale examines the frequency of child and parent behaviors on a Likert scale (1=never and 5=always) and whether or not each item is a problem with "yes" or "no".
Mediation of Children's Media Use | Baseline and at 3 months
  A 16-item parent report of frequency of mediation of children's media use on a Likert scale (1=never and 5=always).
Parent Self-Efficacy | Baseline and at 3 months
  Uses a valid 9-item survey, grouping parents into 3 categories (0-<1.5 not at all/slightly confident; 1.5 - <2.5 very confident; 2.5 - 3 extremely confident).
Parent Nutrition Attitudes | Baseline and at 3 months
  Attitudes of parents toward healthy eating. Measured using an 8-item measure, scored on a range of -2 to +2, with positive scores corresponding with positive attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Gibbs, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States